CLINICAL TRIAL: NCT05617053
Title: DIRECTIONAL ATHERECTOMY WITH ANTIRESTENOTIC THERAPY vs PTA/SUPERA STENTING FOR POPLITEAL ARTERY ATHEROSCLEROTIC LESIONS: A CASE-MATCH PROPENSITY STUDY
Brief Title: DAART vs PTA/SUPERA STENTING FOR POPLITEAL ARTERY LESIONS
Status: Completed | Type: Observational
Sponsor: Vascular Investigation Network Spanish Society for Angiology and Vascular Surgery (Network)
Responsible Party: Principal Investigator, Enrique M. San Norberto, MD, PhD, MSc, MPGCert, Vascular Investigation Network Spanish Society for Angiology and Vascular Surgery
Other Study IDs: PI 22-2967
Record Dates: First submitted 2022-11-01; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Popliteal Artery Stenosis; Atheroma
Keywords: Popliteal artery; Drug-coated balloon; Supera stent; Directional atherectomy
MeSH Terms: conditions — Plaque, Atherosclerotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DAART: Popliteal artery lesion treated by directional atherectomy with anti-restenotic therapy for the treatment of popliteal atherosclerotic lesions.
  Interventions: Device: DAART
- ATP/Supera stenting: Angioplasty and Supera stent implantation for the treatment of popliteal atherosclerotic lesions.
  Interventions: Device: ATP/Supera stenting

INTERVENTIONS:
Device: DAART
  Groups: DAART
Device: ATP/Supera stenting
  Groups: ATP/Supera stenting

SUMMARY:
The purpose of this study was to compare the results of directional atherectomy with antirestenotic therapy (DAART technique) and angioplasty/Supera stenting for the treatment of popliteal atherectomy lesions.

DETAILED DESCRIPTION:
Atherectomy offers a way to improve the chances to avoid stent placement, although it did not show superiority in terms of vessel patency or limb salvage compared with POBA. Nevertheless, atherectomy can modify the plaque morphology and the mechanical properties of the baseline disease, which allows better drug penetration and diffusion into the vessel wall.

Moreover, the combination of directional atherectomy devices and drug coated balloons (directional atherectomy with antirestenotic therapy, DAART), theoretically might further improve the clinical outcomes of drug coated angioplasty. The "leave nothing behind" strategies have gained support among interventionalist. Many studies claim that atherectomy improves results when combined with adjunctive DCB.

The Supera stent, when compared with other self-expanding nitinol stents, has proven to deforms less with knee flexion and exhibits less strain. It mimics the natura structure and movement of the anatomy and optimizes luminal gain maintaining a round open lumen in challenging anatomies, as the popliteal artery. Mechanical scaffolding is often required owing to elastic recoil and flow-limiting dissections in complex popliteal lesions.

The purpose to this study was to retrospectively evaluate the efficacy of both techniques for endovascular treatment of atherosclerotic lesions of the popliteal artery.

ELIGIBILITY:
Inclusion Criteria:

* patients with lifestyle limiting intermittent claudication ischemic rest pain, ischemic ulcers or gangrene (Rutherford class 3 to 6) who presented atherosclerotic lesions in the popliteal artery undergoing endovascular treatment by DAART of PTA/Supera stenting and at least a 12-months of follow-up

Exclusion Criteria:

* Exclusion criteria were patients who could not receive antiplatelet or anticoagulation therapies. Other exclusion criteria were patients with aneurysm of the ipsilateral superficial femoral artery or popliteal artery, acute thrombus, unsalvageable limb, very limited life-expectancy or with doubts in their willingness or capability to allow follow-up examinations.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with lifestyle limiting intermittent claudication, ischemic rest pain, ischemic ulcers or gangrene (Rutherford class 3 to 6) who presented atherosclerotic lesions in the popliteal artery undergoing endovascular treatment by DAART of PTA/Supera stenting and at least a 12-months of follow-up
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Primary latency 12-months | 12 months
  primary patency at 12-months follow-up, defined as absence of binary restenosis or reocclusion on duplex ultrasound examination without repeat target lesion interventions

SECONDARY OUTCOMES:
Secondary Patency | 12-months
  Secondary patency was defined as requiring a secondary intervention to restore patency after occlusion of the treated segment
Mortality | 12-months
  Patients dead all-cause during follow-up
Amputation rate | 12-months
  Patients with minor or mayor amputation during follow-up
Clinical status | 12-months
  Rutherford classification clinical scale after 12-month follow-up
ABI measurement | 12-months
  Ankle/Brachial index measurement.
Stent fracture | 12-months
  Stent fracture and implantation defects were assessed by high-resolution radiographic imaging performed on the stents of every limb
Primary-assisted patency | 12-months
  Primary assisted patency was defined as a patent popliteal segment that underwent further intervention within the inflow, treated vessel segment, or outflow of the treated vessel segment to improve patency

IPD SHARING:
Plan to Share IPD: No